CLINICAL TRIAL: NCT00930579
Title: Phase II Pre-Surgical Intervention Study for Evaluating the Effect of Metformin on Breast Cancer Proliferation
Brief Title: Pre-Surgical Study: Effect of Metformin on Breast Cancer Proliferation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD6525
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metformin
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Women with newly diagnosed early invasive breast cancer will receive Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 1500 mg per day, divided 500 mg in the morning and 1000 mg in the evening, for at least two weeks prior to surgery
  Other Names: Metformin hydrochloride

SUMMARY:
The purpose of this pilot study is to use a pre surgical intervention model to evaluate the biologic effects of metformin in women with newly diagnosed early invasive breast cancer. Metformin is a drug commonly used to treat patients with diabetes. This model will be used to evaluate the effects of metformin.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer and the second leading cause of cancer death among women in the United States. Several epidemiologic studies have found an increased risk of breast cancer in women with type 2 diabetes. This association appears to be mediated by a state of hyperinsulinemia and insulin resistance. Population based studies have also found a decreased risk of cancer in diabetic patients taking metformin, an oral biguanide derivative. Proposed mechanisms include its effect on lowering serum insulin levels as well as modulation of cellular signaling pathways which inhibit tumor cellular proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed operable invasive breast cancer or ductal carcinoma in situ (DCIS) who undergo core needle biopsy followed by surgical excision at least 2 weeks after enrollment
* Body mass index > 25
* Age ≥ 21 years
* No prior chemotherapy, radiation therapy, or surgery within 6 months of study entry
* Signed informed consent

Exclusion Criteria:

* History of diabetes mellitus requiring medical therapy
* Treatment with other investigational drugs within 6 months of study entry
* Significant renal impairment with a creatinine > 1.4 mg/dl
* Other serious intercurrent medical illness

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2012-05-10 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn L Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalinsky K, Zheng T, Hibshoosh H, Du X, Mundi P, Yang J, Refice S, Feldman SM, Taback B, Connolly E, Crew KD, Maurer MA, Hershman DL. Proteomic modulation in breast tumors after metformin exposure: results from a "window of opportunity" trial. Clin Transl Oncol. 2017 Feb;19(2):180-188. doi: 10.1007/s12094-016-1521-1. Epub 2016 Jun 15. PMID 27305912
- [Derived] Kalinsky K, Crew KD, Refice S, Xiao T, Wang A, Feldman SM, Taback B, Ahmad A, Cremers S, Hibshoosh H, Maurer M, Hershman DL. Presurgical trial of metformin in overweight and obese patients with newly diagnosed breast cancer. Cancer Invest. 2014 May;32(4):150-7. doi: 10.3109/07357907.2014.889706. Epub 2014 Mar 7. PMID 24605899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigator conducted an open-label, single-arm, presurgical trial with metformin at Columbia University Medical Center (CUMC) in New York, New York. Between October 2009 and August 2011.
Groups:
- Metformin: Women with newly diagnosed early invasive breast cancer received doses of the study drug, Metformin, prior to their scheduled surgery. Participants received 1500mg of metformin per day - 500mg in the morning, and 1000mg in the evening.
Period: Overall Study
Arm/Group | Metformin
Started | 35
Completed | 33
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Discontinued due to rescheduled surgery | 1

BASELINE CHARACTERISTICS:
Population: Of the 35 patients enrolled, 33 completed the trial and were considered evaluable. Patients were evaluable if they had sufficient pre and post treatment tumor tissue for analysis, and demonstrated at least 75% compliance with metformin, as measured by weekly telephone interviews and pill counts.
Groups:
- Metformin: Women with newly diagnosed early invasive breast cancer received doses of the study drug, Metformin, for at least two weeks before their scheduled surgery. Participants received 1500mg of metformin per day- 500mg in the morning, and 1000mg in the evening.
Arm/Group | Metformin
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 28
  Non-Hispanic White | 2
  Non-Hispanic Black | 2
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Tumor Proliferation in Tumor Specimens
Description: This outcome measure examines the changes in tumor proliferation as measured by the amount of Ki-67 protein in the tumor.
Time Frame: Baseline, up to 4 weeks
Population: Of the evaluable metformin-treated patients, 33 participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of ki-67 positive cells
Groups:
- Metformin: Women with newly diagnosed early invasive breast cancer received doses of the study drug, Metformin, for at least two weeks prior to surgery. Participants received 1500 mg of Metformin per day- 500mg in the morning, and 1000 mg in the evening.
Arm/Group | Metformin
Number analyzed (Participants) | 33
percentage of ki-67 positive cells
  Premetformin Tumor Sample | 2.17 (1.60)
  Post Metformin Tumor Sample | 2.165 (1.67)
Statistical Analysis 1: Comparison: Metformin; Null hypothesis: there will be no statistically significant change between the amount of Ki-67 (protein involved in cell proliferation) in participants' tumor cells before and after taking the prescribed dose of Metformin, as measured at the 5% significance level; Test type: Other — This study used two-sided t-tests to compare changes within group- before and after metformin treatment; p = 0.98, paired t-test; Mean Difference (Final Values) = -0.006

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, is the same as the ClinicalTrials.gov definitions.
Arm/Group | Metformin
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 29/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=33)
Diarrhea (Gastrointestinal disorders) | 21 — Grade 1
Diarrhea (Gastrointestinal disorders) | 5 — Grade 2
Diarrhea (Gastrointestinal disorders) | 3 — Grade 3
Flatulence (Gastrointestinal disorders) | 15 — Grade 1
Nausea (Gastrointestinal disorders) | 11 — Grade 1
Anorexia (Metabolism and nutrition disorders) | 10 — Grade 1
Fatigue (General disorders) | 10 — Grade 1
Dizziness (Nervous system disorders) | 8 — Grade 1
Headache (Nervous system disorders) | 8 — Grade 1
Abdominal Distension (Gastrointestinal disorders) | 7 — Grade 1
Abdominal Pain (Gastrointestinal disorders) | 7 — Grade 1
Taste Alteration (Nervous system disorders) | 6 — Grade 1
Dry Mouth (Investigations) | 5 — Grade 1
Constipation (Gastrointestinal disorders) | 4 — Grade 1
Rash (Skin and subcutaneous tissue disorders) | 4 — Grade 1
Heartburn (Investigations) | 3 — Grade 1
Vomiting (Gastrointestinal disorders) | 3 — Grade 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 — Grade 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes